CLINICAL TRIAL: NCT06516406
Title: Ruxolitinib in Primary Myelofibrosis and Secondary to Essential Thrombocythemia or Polycythemia Vera
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RUX-MF
Record Dates: First submitted 2023-10-05; First posted 2024-07-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-02

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Secondary Myelofibrosis
Keywords: Safety; Efficacy
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is observational multicenter retrospective and prospective cohort study of patients with primary or secondary myelofibrosis who have initiated therapy with ruxolitinib, prescribed as part of the normal course of care and completely independent of study participation. The primary purpose is to determine the impact of clinical and laboratory characteristics of myelofibrosis on the prognosis of patients treated with ruxolitinib, understood as long-term survival.

DETAILED DESCRIPTION:
The study is observational multicenter retrospective and prospective cohort study of patients with primary or secondary myelofibrosis who have initiated therapy with ruxolitinib, prescribed as part of the normal course of care and completely independent of study participation. Laboratory tests and histological, cytogenetic, molecular, and radiological investigations performed by the patient and collected for study will be conducted in accordance with clinical practice, independent of the patient's participation in the study. In particular. data on systemic symptoms and splenomegaly will be collected at diagnosis and disease reassessments performed in the context of normal clinical practice. The minimum planned duration of individual patient observation is 3 months and the planned duration of the study is 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients diagnosed with Primary Myelofibrosis or secondary to Essential Thrombocythemia/Polycythemia vera who are being treated or have been treated with ruxolitinib therapy in accordance with normal clinical practice.
* Availability of data on clinical history prior to initiation of Ruxolitinib therapy
* Obtaining informed consent for data collection and processing

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is observational multicenter retrospective and prospective cohort will be offered consecutively to any patient with primary or secondary myelofibrosis who has initiated therapy with ruxolitinib, prescribed as part of the normal course of care and completely independent of study participation. The study will be conducted in the study-participating OUs of Hematology, and an estimated total of 1015 patients who initiated therapy with Ruxolitinib between 2008 and the end of the study are expected to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1055 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Long Term Survival | 10 years
  To determine the impact of clinical and laboratory characteristics of myelofibrosis on the prognosis of patients treated with ruxolitinib, in terms of long-term survival.

SECONDARY OUTCOMES:
Significance of peripheral blasts | 10 years
  To assess correlations between amount of peripheral blasts and response to treatment, leukaemic transformation, drug withdrawal and survival.
Prognostic value of High Molecular Risk (HMR) mutations. | 10 years
  To assess the prognostic value of HMRs (via NGS) in MF patients treated with ruxolitinib and to develop a prognostic model that can be applied to patients before and during ruxolitinib therapy.
To validate the use of the MTSS score | 10 years
  To validate the use of the MTSS score to assess post-ASCT survival of patients with MF
Incidence of adverse events | 10 years
  To assess the incidence of adverse events in patients with myelofibrosis treated with ruxolitinib: thrombosis, haemorrhage, second neoplasms, blastic evolution.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 10 years
  To assess the toxicity of ruxolitinib therapy in the total cohort

CONTACTS AND LOCATIONS:
Locations (26):
- Italy (26):
  - Azienda Ospedaliera Annunziata, Cosenza, Calabria
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli", Reggio Calabria, Calabria
  - Università degli Studi di Napoli Federico II U.O.C. di Ematologia e Trapianti di midollo, Napoli, Campania
  - IRCCS Policlinico Sant'Orsola, Bologna, Emilia-Romagna
  - Università degli studi di Ferrara - Nuovo Polo Ospedaliero di Cona - A.O.U. Arcispedale S. Anna, Ferrara, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Emilia-Romagna
  - AUSL di Piacenza - Palazzine Medicine Specialistiche, Piacenza, Emilia-Romagna
  - Dipartimento Oncoematologico - AUSL della Romagna, Ravenna, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - A.O.U. Integrata di Udine, Udine, Friuli Venezia Giulia
  - A.O.U. Policlinico Umberto I - Università degli Studi di Roma "La Sapienza", Rome, Lazio
  - Ospedale S. Eugenio, Rome, Lazio
  - Ospedale Belcolle, Viterbo, Lazio
  - IRCCS Azienda Ospedaliera Universitaria "San Martino" - IST, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Ospedale San Luigi Gonzaga - Regione Gonzole, Turin, Piedmont
  - Department of Oncology, University of Torino, Turin, Piedmont
  - Città della Salute e della Scienza, Turin, Piedmont
  - A. O. Ordine Mauriziano di Torino, Turin, Piedmont
  - Ospedale "A. Businco" - Dipartimento Scienze Mediche e Sanità Pubblica Università degli Studi di Cagliari, Cagliari, Sardinia
  - A.O.U. "Policlinico-V. Emanuele"- P.O. Ferrarotto, Catania, Sicily
  - A.O. Ospedali Riuniti Marche Nord - Presidio Ospedaliero San Salvatore, Pesaro, The Marches
  - Policlinico S.Maria alle Scotte, Siena, Tuscany
  - AOU di Padova, Padua, Veneto
  - A.O.U. Integrata Verona, Verona, Veneto